CLINICAL TRIAL: NCT03376620
Title: Role of Topical Putrescine (Fibrostat) in 10%Urea (TFU) for Prevention of Hypertrophic Scars in Mammoplasty Patients
Brief Title: Role of Topical Putrescine (Fibrostat) for Prevention of Hypertrophic Scars in Mammoplasty Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B2008:134
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2017-12-20 (Actual); Status verified 2017-11

CONDITIONS: Hypertrophic Scar
Keywords: Prevention of hypertrophic scar
MeSH Terms: conditions — Cicatrix, Hypertrophic | interventions — Putrescine

STUDY DESIGN:
Intervention Model Description: Double-Blind Randomized Controlled Trial; Patient as their own control
Who Masked: Participant, Investigator
Masking Description: Label number coded by manufacturer and released after blinding period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10% Urea cream (Sham Comparator): Opposite breast scars treated OD at hs simultaneously using sham 10% Urea cream
  Interventions: Drug: 10% Urea cream
- Active cream with 1,4 diaminobutane (Active Comparator): Other breast scar treated daily with active cream with 1,4 diaminobutane topically OD at hs
  Interventions: Drug: 1,4-Diaminobutane

INTERVENTIONS:
Drug: 1,4-Diaminobutane — Daily application to surgical breast scars of 1,4 diaminobutane on the active side
  Other Names: Fibrostat
  Arms: Active cream with 1,4 diaminobutane
Drug: 10% Urea cream — Daily application to surgical breast scars of 10% Urea cream on the sham side
  Arms: 10% Urea cream

SUMMARY:
Linked to previous Clinical Trial E92:069 in which biochemical effect of 1,4 diaminobutane was studied in human scar harvested at revision surgery after a 12 week application. Analytical data was collected in this phase of the work completed in 1999. This was then followed by clinical correlation in a scar prevention model with topical application of 1,4 diaminobutane for 12 weeks and measuring duredness , as well photographic and POSAS score data for quality of scar formation.

DETAILED DESCRIPTION:
In this study, patients were "randomized" into one of 2 study groups described below. They agreed to being treated on the right side or the left with active agent, while the other side was to receive inactive cream. The active molecule is called Fibrostat or 1,4 diaminobutane and is a naturally occurring inhibitor of scar formation. The inactive jar contains the vehicle alone without Fibrostat.

The patients received both cream types to be applied to the appropriate side assigned by the randomization process, one numbered jar each per breast in the order and amount as explained in detail by the patient educator. The cream was applied daily and in the same order, one jar for the right and the other jar for the left consistently. The randomization was performed at the factory with an assigned number recorded on each jar and the jar contents listed and recorded with its assigned number. Each jar of active cream is randomly assigned with another jar of inactive cream to form a pair which were both given to the patient. The cream in both jars looks and smells the same. Neither the patient nor the study doctor knew which breast as receiving the active agent. In an emergency, this information was to be made available.

Participation in the study was for 12 weeks. the patients were seen for photos and scar testing using a painless surface testing device called a Rex® durometer at 1, 3, 6, and 12 weeks post op.

The researcher could decide to take patients off this study if a patient were to develop a rash during the run-in period of 1 week from the cream on either side.

The patients could stop participating at any time. However, this was usually accompanied by a valid reason such as lack of transportation to regular follow up appointments. No serious effects were seen and the only patients to stop participation in the study except 1 which was lost to follow-up could be accounted for. The results were revealed to patients at the completion of the 12 week trial.

ELIGIBILITY:
Inclusion Criteria: Undergoing breast reduction surgery -

Exclusion Criteria: Not pregnant or lactating

-

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-09-02 (Actual); Primary Completion 2013-08-13 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Duredness of scar at post treatment time frame for active versus control breast | 12 weeks
  Surface deformational force in grams of scar tissue in each of the treated breasts

SECONDARY OUTCOMES:
Patient Observer Objective Scar Assessment Scale ratings | at least one year post operatively
  Validated scale of scar outcome based on seven parameters graded on a scale of 1-10 ranked lowest to highest in severity. Patient was the "observer" in this study making subjective parameters listed such as pain and itch a direct patient correlate rather than one recorded by a second-person observation.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dolynchuk KN, Tredget EE. A Preliminary Report of the Biochemical and Clinical Effects of 1,4-Diaminobutane on Prevention of Human Hypertrophic Scars. Plast Reconstr Surg. 2020 Jan;145(1):76e-84e. doi: 10.1097/PRS.0000000000006413. PMID 31881614